CLINICAL TRIAL: NCT03264131
Title: Brentuximab Vedotin With Cyclophosphamide, Doxorubicin, Etoposide, and Prednisone (BV-CHEP) for the Treatment of Adult T-Cell Leukemia/Lymphoma: A Pilot Study of the Rare Lymphoma Working Group
Brief Title: BV-CHEP Chemotherapy for Adult T-cell Leukemia or Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1637
Record Dates: First submitted 2017-08-15; First posted 2017-08-28 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma; Adult T-Cell Leukemia/Lymphoma; Lymphatic Diseases
Keywords: Brentuximab Vedotin; Adcetris; Lymphoma; Leukemia; CD30
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphatic Diseases; Leukemia | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label, Multicenter, Single-Arm (Experimental): This is a single-arm intervention where patients will receive concurrent therapy with BV+CHEP [(brentuximab vedotin; 1.8 mg/kg IV, on D1 every 21 days) (cyclophosphamide 750 mg/m^2 on D1; doxorubicin 50 mg/m^2 on D1, etoposide 100 mg/m^2 IV infusion on D1-3; prednisone 100 mg orally once daily on D1-5; cycle length every 21 days)] for 2 to 6 cycles of induction therapy. After 6 cycles of BV + CHEP, responders (CR, PR or SD) who are not eligible for BMT and have CD30-positive ATLL will continue maintenance therapy with BV alone (1.8 mg/kg IV, every 21 days) until disease progression, withdrawal due to toxicity or death.
  Interventions: Drug: Brentuximab Vedotin; Drug: CHEP

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab Vedotin will be given at 1.8 mg/kg IV over approximately 30 minutes on D1 every 21 days for 2-6 cycles. Responders (CR, PR or SD) who are not eligible for bone marrow transplant (BMT) and have CD30-positive ATLL will continue maintenance therapy with BV alone (1.8 mg/kg IV for approximately 30 minutes, every 21 days).
Drug: CHEP — Cyclophosphamide- 750 mg/m^2 IV over approximately 1 hour on D1 every 21 days for 2-6 cycles
  Doxorubicin- 50 mg/m^2 IV over approximately 3-5 minutes on D1 every 21 days for 2-6 cycles.
  Etoposide - 100 mg/m^2 IV over approximately 1 hour each day for 3 days every 21 days for 2-6 cycles.
  Prednisone - 100 mg, orally once daily for 5 days every 21 days for 2-6 cycles.

SUMMARY:
Adult T-cell leukemia/lymphoma (ATLL) is a rare form of cancer found mostly among people from the Caribbean islands, Western Africa, Brazil, Iran, and Japan. Most cases of this disease in the United States occur along the East Coast due to emigration from the Caribbean islands. There is currently no standard treatment for ATLL. Research shows that patients who go into first time remission (respond completely or partially to treatment) and have a bone marrow transplant have the best outcomes. Traditional chemotherapy treatments have generally not worked well in patients with ATLL. Additionally, not all patients will be eligible for a bone marrow transplant.

The purpose of this study is to see how well individuals with ATLL respond to an investigational cancer treatment. This investigational treatment combines a drug called brentuximab vedotin with a standard chemotherapy treatment made up of cyclophosphamide, doxorubicin, etoposide, and prednisone. This treatment is considered investigational because it is not approved by the United States Food and Drug Administration (FDA) for the treatment of ATLL.

Brentuximab vedotin, also known as Adcetris, is approved by the United States Food and Drug Administration (FDA) for treatment of certain types of lymphomas, including peripheral T-cell lymphomas when combined with cyclophosphamide, doxorubicin, and prednisone in patients whose cancer cells express a type of marker called CD30.

Brentuximab vedotin is an antibody that also has a chemotherapy drug attached to it. Antibodies are proteins that are part of the immune system. They can stick to and attack specific targets on cancer cells. The antibody part of brentuximab vedotin sticks to a target called cluster of differentiation 30 (CD30) that is located on the outside of the cancer cells. Normal cells have little or no CD30 on their surface. ATLL cancer cells often have a larger amount of CD30 on their surface than normal cells. However, CD30 is found in different amounts on ATLL cancer cells. This study will also test the amount of CD30 found on each participant's cancer cells. Researchers will be looking to see if the response to the study treatment varies based on the amount of CD30 found on the outside participants' cancer cells.

In another study, brentuximab vedotin was combined in another study with cyclophosphamide, doxorubicin, and prednisone. The study included patients with various types of T-cell lymphomas. Two of the patients enrolled in that study had ATLL. Both had a complete response (no evidence of disease). The researchers in this study (LCCC 1637) have added etoposide to the combination of brentuximab vedotin with cyclophosphamide, doxorubicin, and prednisone. They predict that the addition of etoposide will improve patient outcomes. Research shows that etoposide helps improve outcomes in patients with certain types of T-cell lymphomas who undergo chemotherapy treatment. This investigational combination of brentuximab vedotin with cyclophosphamide, doxorubicin, etoposide, and prednisone is called BV-CHEP.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Objective To define the proportion of subjects with CR after 4-6 cycles of brentuximab vedotin in combination with cyclophosphamide, doxorubicin, etoposide, and prednisone (BV-CHEP) in the treatment of adult T-cell leukemia/lymphoma.

Secondary Objectives

To estimate the overall response rate (ORR) with 4-6 cycles of BV-CHEP therapy in patients with adult T-cell leukemia/lymphoma.

To determine progression-free survival (PFS) for BV-CHEP in patients with adult T-cell leukemia/lymphoma who received or did not receive BV maintenance.

To determine duration of response to BV-CHEP in patients with adult T-cell leukemia/lymphoma who received or did not receive BV maintenance.

To determine overall survival (OS) of patients with adult T-cell leukemia/lymphoma treated with BV-CHEP who received or did not receive BV maintenance therapy.

To evaluate the toxicity and tolerability of BV-CHEP and BV maintenance therapy via the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03).

*Note: After completion or withdrawal from BV-CHEP therapy, patients will segregate into one of the following groups: 1) those who progressed on BV-CHEP; 2) those who completed 4-6 cycles of BV-CHEP and went on to allogeneic transplant; 3) those who completed 6 cycles of BV-CHEP but were CD30 negative and ineligible for maintenance therapy; and 4) those who completed 6 cycles of BV-CHEP, were CD30 positive, but continued study treatment on BV in the maintenance phase of the study.

ENDPOINTS

Primary Endpoint

Criteria for CR after 4-6 cycles of BV-CHEP will be based on the International Workshop to standardize response criteria for malignant lymphomas (ie, Lugano Criteria per Cheson, et al. J Clin Oncol. 2014;32(27):3059-68).

Secondary Endpoints

Criteria for overall response will be based on the International Workshop to standardize response criteria for malignant lymphomas (ie, Lugano Criteria per Cheson, et al. J Clin Oncol. 2014;32(27):3059-68).

PFS is defined as time from D1 of treatment until disease progression (based on Lugano criteria) or death from any cause.

Duration of response is defined as the time from documentation of tumor response per Lugano criteria to disease progression

OS is defined as the time from D1 of treatment until death from any cause

Toxicity and tolerability of therapy will be assessed via the NCI CTCAE v4.03

TREATMENT INFORMATION

Patients will undergo screening to see if they are eligible. If eligible, participants will start by receiving 2 cycles of BV-CHEP (cycles 1 and 2). After 2 cycles of BV-CHEP, participants will have a positron emission tomography/computed tomography (PET/CT) or a CT scan to assess their disease. If the scan shows the cancer has stayed the same or gotten better, participants may continue taking BV-CHEP for two more cycles (cycle 3 and 4). If, at any time during study treatment, a participant's disease gets worse, the participant will end study treatment and other treatment options will be discussed with you.

If a participant continues on BV-CHEP, at the beginning of cycle 5, the participant will have a PET/CT scan. If the cancer has gotten better and the participant is eligible for a bone marrow transplant, he/she will have the transplant. If the participant is not eligible for a bone marrow transplant and the cancer has stayed the same or gotten better, the participant may continue on BV-CHEP for two more cycles (cycles 5 and 6).

At the end of cycle 6 of BV-CHEP, participants will have another PET/CT scan. If the scan shows the cancer has gotten better and the participant is eligible for a bone marrow transplant, he/she will have the transplant. If a participant is not eligible for a bone marrow transplant and his/her cancer cells did not test positive for CD30, the participant will end study treatment. The study doctor will discuss other treatment options that are not part of this study with the participant.

Participants may continue on brentuximab vedotin alone as maintenance therapy if:

* They are not eligible for a bone marrow transplant,
* Their cancer cells tested positive for CD30, and
* Their cancer has not gotten worse after taking BV-CHEP.

Participants will be removed from BV maintenance therapy if their cancer get worse.

DURATION OF THERAPY Therapy in LCCC 1637 involves up to 6 cycles of treatment with brentuximab vedotin (BV) with a chemotherapy treatment made up of cyclophosphamide, doxorubicin, etoposide, and prednisone (CHEP). Each cycle is 21 days long. Participants may continue on BV alone as maintenance therapy after 6 cycles of BV-CHEP if they meet the requirements outlined above. Each cycles of BV maintenance therapy is 21-day long. BV maintenance therapy may continue until a participant's disease progresses.

DURATION OF FOLLOW-UP PERIOD Participants will be followed for survival for up to 5 years. They will also have a PET/CT or CT scan and a blood test every 6 months for 2 years after study treatment ends.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to participate in this study:

1. Informed consent and HIPAA authorization for release of personal health information obtained.
2. Age ≥ 18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
4. Histological confirmation of biopsy-proven peripheral T-cell leukemia/lymphoma consistent with ATLL

   * Included subtypes will be: acute, lymphomatous, and chronic unfavorable. Chronic unfavorable is defined as the chronic variant with at least one of the following: lactate dehydrogenase (LDH)>upper limit of normal (ULN), blood urea nitrogen (BUN)>ULN, Albumin<lower limit of normal (LLN)
   * Positive human T-lymphotropic virus-1 (HTLV-1) antibody testing with confirmatory testing via Western blot, enzyme-linked immunosorbent assay (ELISA), or molecular testing (PCR).
5. Documented negative serologic testing for human immunodeficiency virus (HIV).
6. If positive for HBV exposure or prior infection, can continue to participate in trial with prophylactic entecavir (for HBV). If positive for hepatitis c virus (HCV) exposure or active infection, can participate in trial with monitoring for liver function abnormalities.
7. Demonstrate adequate organ function as defined below; all screening labs to be obtained within three days prior to study treatment.

   System: Renal -Calculated creatinine clearance

   Laboratory Value: ≥ 30 mL/min using the Cockcroft-Gault formula for subjects with creatinine levels > 2.0 x institutional ULN

   System: Hepatic - Bilirubin

   Laboratory Value: ≤ 3.0 mg/dL

   System: Hepatic - Aspartate aminotransferase (AST)

   Laboratory Value: ≤ 2.5 × ULN

   System: Hepatic - Alanine aminotransferase (ALT)

   Laboratory Value: ≤ 2.5 × ULN
8. Females of childbearing potential must have a negative serum pregnancy test within three days (72 hours) prior to initiating study treatment. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
9. Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 24 weeks (6 months) after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets <1% failure rate for protection from pregnancy in the product label.
10. Male patients with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 24 weeks (6 months) after the last dose of study therapy.
11. As determined by the enrolling physician or protocol designee, willingness and ability of the subject to understand and comply with study procedures
12. Prior Treatment: Previously untreated or has received a maximum of one cycle of any combination chemotherapy (e.g. cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP), CHOEP, DA-EPOCH, doxorubicin, cyclophosphamide, cytarabine, vincristine, methotrexate/Etoposide, ifosfamide, cytarabine, methotrexate (CODOX-M/IVAC), HyperCVAD) within 4 weeks of signing the main consent form. Additionally, a patient may have taken antiretroviral therapy (e.g. azidothymidine (AZT) and/or IFN) at any time prior to study enrollment
13. CD30 expression determined by flow cytometry or IHC. NOTE: If CD30 testing was previously done on the biopsy sample from diagnosis, this information will be collected. If CD30 testing was not done, an archival sample from the biopsy used for diagnosis will be requested and tested for CD30. CD30 testing will also be done on the bone marrow tissue collected from the bone marrow exam. If we are unable to obtain an archival sample or if the bone marrow exam is negative, a new biopsy will be performed to confirm the diagnosis and test for CD30.

Exclusion Criteria:

Subjects who meet any of the following criteria should be excluded from study participation:

1. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
2. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
3. Previous exposure to brentuximab vedotin (BV).
4. History of allergic response to BV-CHEP or its components or to any of the required prophylactic medications or reasonable alternatives.
5. Symptomatic cardiac disease including ventricular dysfunction, left ventricular ejection fraction < 40%, symptomatic coronary artery disease or symptomatic arrhythmias
6. Subjects with severe hepatic insufficiency Child-Pugh Score > 6
7. Subjects with severe renal impairment (i.e., creatinine clearance ≤ 30 mL/min; see Appendix B - Renal Impairment Guidelines).
8. Exclude patients with pre-existing neuropathy grade 2 or higher.
9. Patients receiving prohibited medications listed in the patient handout provided in 11.4 Appendix D: Prohibited Medications or Those to be used with Caution (ie, ketoconazole, itraconazole, ritonavir, macrolide antibiotics, erythromycin phenytoin, phenobarbital, carbamazepine, and valproic acid).
10. Patients with a parenchymal brain lesion thought to be consistent with active lymphoma on screening CT/MRI. Of note, patients with cerebrospinal fluid (CSF) involvement alone are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2028-12-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dittus Christopher, DO, MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (4):
- United States (4):
  - South Broward/Memorial Healthcare System, Hollywood, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Lineberger Comprehensive Cancer Center at the University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — https://unclineberger.org/research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study between 10/11/2018 - 06/22/2022 at four cancer centers in the United States.
Pre-assignment Details: A total of sixteen eligible participants consented and started to the study.
Groups:
- Open-label, Multicenter, Single-Arm: This is a single-arm intervention where patients will receive concurrent therapy with BV+CHEP [(brentuximab vedotin; 1.8 mg/kg IV, on D1 every 21 days) (cyclophosphamide 750 mg/m^2 on D1; doxorubicin 50 mg/m^2 on D1, etoposide 100 mg/m^2 IV infusion on D1-3; prednisone 100 mg orally once daily on D1-5; cycle length every 21 days)] for 2 to 6 cycles of induction therapy. After 6 cycles of BV + CHEP, responders (CR, PR or SD) who are not eligible for BMT and have CD30-positive ATLL will continue maintenance therapy with BV alone (1.8 mg/kg IV, every 21 days) until disease progression, withdrawal due to toxicity or death.
  Brentuximab Vedotin: Brentuximab Vedotin will be given at 1.8 mg/kg IV over approximately 30 minutes on D1 every 21 days for 2-6 cycles. Responders (CR, PR or SD) who are not eligible for bone marrow transplant (BMT) and have CD30-positive ATLL will continue maintenance therapy with BV alone (1.8 mg/kg IV for approximately 30 minutes, every 21 days).
  CHEP: Cyclophosphamide- 750 mg/m^2 IV over approximately 1 hour on D1 every 21 days for 2-6 cycles
  Doxorubicin- 50 mg/m^2 IV over approximately 3-5 minutes on D1 every 21 days for 2-6 cycles.
  Etoposide - 100 mg/m^2 IV over approximately 1 hour each day for 3 days every 21 days for 2-6 cycles.
  Prednisone - 100 mg, orally once daily for 5 days every 21 days for 2-6 cycles.
Period: Overall Study
Arm/Group | Open-label, Multicenter, Single-Arm
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants consented and started the study.
Arm/Group | Open-label, Multicenter, Single-Arm
Number analyzed (Participants) | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [43.75 to 65.50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate After 2-6 Cycles of Brentuximab Vedotin in Combination With Cyclophosphamide, Doxorubicin, Etoposide, and Prednisone (BV-CHEP)
Description: The response was assessed based on the International Workshop to standardize response criteria for malignant lymphomas (i.e., Lugano Criteria per Cheson, et al. J Clin Oncol. 2014;32(27):3059-68; Complete Response: Positron emission tomography (PET): Complete metabolic response Computerized tomography (CT): Target must regress to ≤ 1.5 cm in the largest transverse diameter (LDi) or no extra lymphatic sites of disease. Partial Response: PET: reduced uptake compared with baseline, and CT: ≥50% decrease in the sum of the products of diameters (SPD).No Response or Stable Disease: No metabolic response on PET or < 50% decrease from baseline in SPD of up to 6 dominant, measurable nodes and extra nodal sites on CT. Progressive Disease: PET: Score 4 or 5 with an increase in the intensity of uptake or CT: an individual node/lesion must be abnormal with LDi > 1.5 cm, increase by ≥ 50% from the cross product of the LDi and shortest axis perpendicular to LDi (SDi).
Time Frame: 18 weeks
Population: Participants started the study and response assessments were completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label, Multicenter, Single-Arm
Number analyzed (Participants) | 16
Participants
  Complete Response | 10
  Partial Response | 4
  Progressive Disease | 2

2. Secondary Outcome: Overall Response Rate (ORR) Associated With 2-6 Cycles of BV-CHEP Therapy in Patients With Adult T-Cell Leukemia/Lymphoma.
Description: ORR will be evaluated as the rate of complete responses (CR) + partial responses (PR) as defined by the International Workshop to standardize response criteria for malignant lymphomas (i.e. Lugano Criteria). Patients with leukemic component to their disease at baseline will be assessed per Adult T-Cell Leukemia/Lymphoma National Comprehensive Cancer Network (NCCN) guidelines version 2.2017
Time Frame: 70 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival (PFS) for BV-CHEP in Patients With Adult T-cell Leukemia/Lymphoma Who Received or Did Not Receive BV Maintenance.
Description: PFS will be assessed from day 1 of treatment until disease progression (based on International Workshop to standardize response criteria for malignant lymphomas (i.e. Lugano Criteria) or death.
Time Frame: 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Response to BV-CHEP in Patients With Adult T-cell Leukemia/Lymphoma Who Received or Did Not Receive BV Maintenance.
Description: Duration of response is defined as the time from documentation of tumor response per Lugano criteria to disease progression. Subjects with a leukemic component to their disease at baseline will have peripheral blood assessed per adult T-cell leukemia/lymphoma NCCN Guidelines version 2.2017
Time Frame: 3 years
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS) of Patients With Adult T-cell Leukemia/Lymphoma Treated With BV-CHEP Who Received or Did Not Receive BV Maintenance Therapy.
Description: Overall survival is defined as the time from day 1 of treatment until death from any cause.
Time Frame: 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Toxicity and Tolerability of BV-CHEP and BV Maintenance Therapy Via National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4)
Description: Toxicity and tolerability of therapy will be assessed via the NCI CTCAE v4.03, a scale from 1-mild to 5-death.
Time Frame: 70 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment. (Up to 14 months)
Description: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03). All hospitalization was graded as SAE per protocol criteria.
Arm/Group | Open-label, Multicenter, Single-Arm
All-Cause Mortality (participants affected / at risk) | 12/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Multicenter, Single-Arm (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Eye pain (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2
pain (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Multicenter, Single-Arm (N=16)
Anemia (Blood and lymphatic system disorders) | 7
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 7
Oral pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 6
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 3
Infections and infestations - Other, specify (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Carbon monoxide diffusing capacity decreased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 4
Lymphocyte count decreased (Investigations) | 3
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Radiculitis (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Cystitis noninfective (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study publication should be a joint publication of all sites. A separate site publication is restricted until 24 months after the study completion or study publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT03264131/Prot_SAP_000.pdf